CLINICAL TRIAL: NCT00787917
Title: An Exploratory, Randomized, Double-blind, Placebo Controlled Study to Assess the Efficacy of Multiple Doses of Omalizumab in Cystic Fibrosis Complicated by Allergic Bronchopulmonary Aspergillosis (ABPA)
Brief Title: An Exploratory Study to Assess Multiple Doses of Omalizumab in Patients With Cystic Fibrosis Complicated by Acute Bronchopulmonary Aspergillosis (ABPA)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIGE025A2437
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Cystic Fibrosis; Allergic Bronchopulmonary Aspergillosis
Keywords: Cystic Fibrosis; Allergic Bronchopulmonary Aspergillosis; omalizumab; oral corticosteroid use; anti-immunoglobulin E
MeSH Terms: conditions — Cystic Fibrosis; Aspergillosis, Allergic Bronchopulmonary | interventions — Omalizumab; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Omalizumab (Experimental): Eligible participants received a maximum dose of 600 mg omalizumab via subcutaneous injection for 6 months in the double-blind phase of the study. The study medication was to be administered at the same time of day. Study medication was injected subcutaneously into the upper arm in the area of the deltoid or to the thigh. A maximum 600 mg dose required 4 injections. All participants who entered the study received itraconazole twice daily, while receiving oral corticosteroids, with a maximum daily dose of 400 mg.
  Participants who completed double-blinded phase, entered open-label treatment period of 6 months and continued the same regimen of omalizumab of double-blinded phase.
  Interventions: Drug: Omalizumab; Drug: Itraconazole
- Placebo (Placebo Comparator): Eligible participants received placebo comparator via subcutaneous injection for 6 months in the double-blind phase of the study. The study medication was to be administered at the same time of day. Study medication was injected subcutaneously into the upper arm in the area of the deltoid or to the thigh. All participants who entered the study received itraconazole twice daily, while on oral corticosteroids, with a maximum daily dose of 400 mg.
  Interventions: Drug: Placebo; Drug: Itraconazole

INTERVENTIONS:
Drug: Omalizumab — Omalizumab subcutaneous injections of 600 mg daily.
  Other Names: Xolair; IGE025
  Arms: Omalizumab
Drug: Placebo — Placebo subcutaneous injections blinded to match experimental arm dosing regimen.
  Arms: Placebo
Drug: Itraconazole — Itraconazole twice daily with a maximum daily dose of 400 mg.
  Other Names: Sporanox

SUMMARY:
This study will evaluate the safety and efficacy of omalizumab for the treatment of Allergic Bronchopulmonary Aspergillosis (ABPA) in patients with Cystic Fibrosis aged 12 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis complicated by Allergic Bronchopulmonary Aspergillosis (ABPA)
* Oral corticosteroid use for ABPA flare
* Age 12 years and older (except for Italy; ≥ 18 years)
* Total serum IgE levels ≥ 500 IU/mL

Exclusion Criteria:

* History of cancer in the last 10 years.
* History of severe allergic reactions
* Pregnant and lactating women
* Prior use of Xolair

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis Investigator Site
Locations (10):
- Novartis Investigator Site, Leuven, Belgium
- Germany (3):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Bonn
  - Novartis Investigator Site, Munich
- Italy (2):
  - Novartis Investigator Site, Milan
  - Novartis Investigator Site, Rome
- Netherlands (2):
  - Novartis Investigator Site, Nijmegen
  - Novartis Investigator Site, Utrecht
- United Kingdom (2):
  - Novartis Investigator Site, Cambridge
  - Novartis Investigator Site, London

REFERENCES:
- [Derived] Beam KT, Coop CA. Steroid sparing effect of omalizumab in seropositive allergic bronchopulmonary aspergillosis. Allergy Rhinol (Providence). 2015 Jan;6(2):143-5. doi: 10.2500/ar.2015.6.0128. PMID 26302738

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab: Eligible participants received a maximum dose of 600 mg omalizumab via subcutaneous injection for 6 months in the double-blind phase of the study. The study medication was to be administered at the same time of day. Study medication was injected subcutaneously into the upper arm in the area of the deltoid or to the thigh. A maximum 600 mg dose required 4 injections. All participants who entered the study received itraconazole twice daily, while receiving oral corticosteroids, with a maximum daily dose of 400 mg.
  Patients completed double-blinded phase, entered open-label treatment period of 6 months and continued the same regimen of omalizumab of double-blinded phase.
Period: Blinded Treatment
Arm/Group | Omalizumab | Placebo
Started | 9 | 5
Completed | 4 | 3
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Administrative problems | 3 | 2
Period: Open Label
Arm/Group | Omalizumab | Placebo
Started | 7 | 0 ("Placebo" was not an arm in open label treatment.)
Completed | 3 | 0
Not Completed | 4 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 0
Not completed — Administrative problems | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 9 | 5 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 21 (4.1) | 28 (9.5) | 23 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline, as Measured by the Percentage of Participants Requiring Rescue With Corticosteroids, and as Measured by the Time to Deviation From the Protocol Prescribed Steroid Tapering Regimen
Time Frame: 6 months of blinded treatment
Population: No statistical analysis was performed due to insufficient study enrollment
Measure: Least Squares Mean (Standard Error); unit: percentage
Groups:
- Omalizumab: Eligible participants received a maximum dose of 600 mg omalizumab via subcutaneous injection for 6 months in the double-blind phase of the study. The study medication was to be administered at the same time of day. Study medication was injected subcutaneously into the upper arm in the area of the deltoid or to the thigh. A maximum 600 mg dose required 4 injections. All participants who entered the study received itraconazole twice daily, while receiving oral corticosteroids, with a maximum daily dose of 400 mg.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Allergic Bronchopulmonary Aspergillosis (ABPA) Exacerbation Rates During Double-blind Treatment Period and Open-label Treatment Period
Time Frame: 6 months, 12 months
Population: No statistical analysis was performed due to insufficient study enrollment
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) From Baseline, Measured at 3 and 6 Months of Treatment
Time Frame: 3 months, 6 months
Population: No statistical analysis was performed due to insufficient study enrollment
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Steroid Free State.
Time Frame: 12 months
Population: No statistical analysis was performed due to insufficient study enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Average Oral Corticosteroid Use.
Time Frame: 6 months, 12 months
Population: No statistical analysis was performed due to insufficient study enrollment
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants Responding to Omalizumab, as Defined by a Reduction in Oral Corticosteroid Dose Use of 50% or More as Compared to Baseline
Time Frame: 6 months, 12 months
Population: No statistical analysis was performed due to insufficient study enrollment
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Blinded Omalizumab: Eligible participants received a maximum dose of 600 mg omalizumab via subcutaneous injection for 6 months in the double-blind phase of the study. The study medication was to be administered at the same time of day. Study medication was injected subcutaneously into the upper arm in the area of the deltoid or to the thigh. A maximum 600 mg dose required 4 injections. All participants who entered the study received itraconazole twice daily, while receiving oral corticosteroids, with a maximum daily dose of 400 mg.
- Open Label Omalizumab: Patients who completed double-blinded phase of the study, enrolled into 6 months open label phase and continued in the same regimen of omalizumab as they were during double-blinded phase. A maximum dose of 600 mg omalizumab via subcutaneous injection for 6 months was to be administered at the same time of day. Study medication was injected subcutaneously into the upper arm in the area of the deltoid or to the thigh. A maximum 600 mg dose required 4 injections. All participants who entered the study received itraconazole twice daily, while receiving oral corticosteroids, with a maximum daily dose of 400 mg.
Arm/Group | Blinded Omalizumab | Placebo | Open Label Omalizumab
Serious Adverse Events (participants affected / at risk) | 6/9 | 1/5 | 4/7
Other Adverse Events (participants affected / at risk) | 9/9 | 5/5 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Omalizumab (N=9) | Placebo (N=5) | Open Label Omalizumab (N=7)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 2 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 5 | 1 | 4
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Omalizumab (N=9) | Placebo (N=5) | Open Label Omalizumab (N=7)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Chills (General disorders) | 0 | 1 | 0
Device occlusion (General disorders) | 1 | 0 | 0
Exercise tolerance decreased (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 3 | 0 | 0
Injection site inflammation (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0
Injection site swelling (General disorders) | 4 | 0 | 0
Injection site warmth (General disorders) | 4 | 0 | 0
Medical device pain (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 2 | 2
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 6 | 4 | 3
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis's agreements with it's investigators vary. However, Novartis does not prohibit any investigator from publishing. Any publication from a single-center site are postponed until the publication of the pooled data ( i.e. data from all sites) in the clinical trial.